CLINICAL TRIAL: NCT01831206
Title: Collagen Cross-linking in Infectious Keratitis Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Ngamjit Kasetsuwan, Associated professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 438/55
Record Dates: First submitted 2013-04-06; First posted 2013-04-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2013-04

CONDITIONS: Infectious Keratitis; Bacterial Keratitis; Fungal Keratitis
Keywords: corneal ulcer; keratitis
MeSH Terms: conditions — Corneal Ulcer; Keratitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collagen cross-linking (Experimental): Collagen cross-linking with standard treatment
  Interventions: Procedure: Collagen cross-linking
- standard treatment (No Intervention): Standard treatment alone

INTERVENTIONS:
Procedure: Collagen cross-linking — Collagen cross-linking arm will receive standard medication for corneal ulcer treatment and corneal collagen cross-linking.
  Standard treatment arm will receive only standard medication.
  Arms: Collagen cross-linking

SUMMARY:
The purpose of this study is to evaluate the efficacy of collagen cross-linking for treatment of infectious keratitis.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of corneal ulcer grade II or III (bacteria or fungal, or presumed bacterial or fungal)
* Age more than 6 year
* Patients can understand and can follow the study protocol

Exclusion Criteria:

* Pregnancy by history or urine test
* Evidence of herpetic keratitis
* Evidence of corneal perforation
* Evidence of autoimmune disease
* Known allergy to study medication

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
decrement of infiltration size | 1 months
  decrement of infiltration size between day0 and day 30

SECONDARY OUTCOMES:
number of participants with adverse events | 1 months
  adverse events after corneal collagen cross-linking (report in descriptive study)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology department, King Chulalongkorn Memorial hospital, Pratumwan, Bangkok, Thailand

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558